CLINICAL TRIAL: NCT06406816
Title: Neoantigen Vaccine Plus Capecitabine as Adjuvant Therapy for Intrahepatic Cholangiocarcinoma After Radical Resection
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yongyi Zeng (Other)
Responsible Party: Sponsor-Investigator, Yongyi Zeng, Director, Meng Chao Hepatobiliary Hospital of Fujian Medical University
Organization: Meng Chao Hepatobiliary Hospital of Fujian Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024_033_01
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoantigen Vaccine plus Capecitabine (Experimental): Neoantigen Vaccine plus Capecitabine for the treatment of high-risk recurrent intrahepatic cholangiocarcinoma
  Interventions: Combination Product: Neoantigen Vaccine plus Capecitabine

INTERVENTIONS:
Combination Product: Neoantigen Vaccine plus Capecitabine — 1. Capecitabine.Twice a day, 30 minutes after breakfast, swallow with water, continue for 2 weeks, then stop for 1 week, constitutes one cycle; three weeks make one cycle, lasting for 8 cycles.
  2. Neoantigen Vaccine . Every 3 weeks, once every 21 days, for 4 to 8 cycles. The injection is administered on the first day after cessation of capecitabine. Treatment can last for up to 6 months without occurrences such as the researcher determining no further clinical benefit, intolerable toxic reactions, initiation of new anti-tumor treatment, withdrawal of informed consent, loss to follow-up, death, or other circumstances specified in the protocol that require treatment termination.

SUMMARY:
This study is a single-arm, open-label, exploratory clinical trial, with the primary objective to evaluate the efficacy and safety of the Neoantigen Vaccine plus capecitabine for the treatment of high-intermediate risk recurrent intrahepatic cholangiocarcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Sign a written informed consent form and be able to comply with the scheduled visits and related procedures as per the protocol;
2. Age ≥18 years and ≤75 years, any gender;
3. Confirmed pathologically as a patient with intrahepatic cholangiocarcinoma;
4. Not receiving neoadjuvant therapy, underwent surgical resection, and pathology confirmed high-risk factors for recurrence: positive margins, lymph node metastasis, vascular invasion, nerve invasion, diameter >5cm, classified as stage IB-IIIB according to AJCC TNM (8th edition, 2017), and have not yet received systemic adjuvant therapy;
5. Child-Pugh score grade A;
6. ECOG score of 0-1;
7. If infected with hepatitis B virus (HBV), such as HBsAg positive, HBV-DNA must be tested and HBV-DNA should be <2000 IU/mL (if the research center uses copy/mL as the detection unit, then it must be <104 copy/mL), and must have received at least 1 week of anti-HBV treatment before the start of the study and willing to undergo antiviral treatment throughout the study period; HCV RNA positive patients must receive antiviral treatment according to the treatment guidelines;
8. The subjects are required to provide fresh or archived tumor tissue samples as requested in the post-operative protocol for use in gene sequencing and peptide gel vaccine preparation;
9. Expected survival period ≥12 weeks;
10. Has sufficient organ and bone marrow function, has not received blood transfusion or hematopoietic growth factor within 14 days before screening. Laboratory test values meet the following requirements, as follows: a. Hematology: Absolute neutrophil count (ANC) ≥1.5×10^9/L; Platelet count (PLT) ≥50×10^9/L; Hemoglobin (HGB) ≥90g/L b. Liver function: Total bilirubin (TBIL) ≤3×upper limit of normal value (ULN); Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) ≤5×ULN; Serum albumin ≥30g/L c. Renal function: Serum creatinine (Cr) ≤1.5×ULN, or for subjects with creatinine >1.5×ULN, creatinine clearance rate (CCr) ≥45 mL/min (Cockcroft-Gault formula); Urine routine results show urine protein <2+; For subjects with urine protein ≥2+ on baseline urine routine testing, 24-hour urine collection should be performed and 24-hour urine protein quantification <1 g d. Coagulation function: International normalized ratio (INR) or APTT ≤1.5×ULN;
11. Fertile women: Must agree to abstain from sexual intercourse (avoid heterosexual intercourse) or use a reliable and effective method of contraception from the start of signing the informed consent form until at least 120 days after the last dose of study drug. Serum HCG test must be negative in the week before treatment; and must be non-lactating. If female patients have menstruated and have not reached postmenopausal status (consecutive absence of menstruation for ≥12 months, no other reason except for menopause), and have not undergone sterilization surgery (such as hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), they are considered fertile;
12. For male subjects with fertile female partners, must agree to abstain from sexual intercourse or use a reliable and effective method of contraception from the start of signing the informed consent form until at least 120 days after the last dose of study drug. Male subjects must also agree not to donate sperm during the same period. Male subjects whose partners are pregnant must use condoms, and no other contraceptive method is necessary

Exclusion Criteria:

1. Pathological diagnosis of hepatocellular carcinoma, mixed hepatocellular carcinoma, hilar cholangiocarcinoma, and gallbladder cancer;
2. Patients with other active malignant tumors other than intrahepatic cholangiocarcinoma within 5 years or simultaneously. Patients with localized tumors that have been cured, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, prostatic carcinoma in situ, cervical carcinoma in situ, breast carcinoma in situ, etc., can be included;
3. Currently with interstitial pneumonia or interstitial lung disease, or with a history of interstitial pneumonia or interstitial lung disease requiring steroid treatment in the past, or other possible interferences with the judgment and treatment of immune-related pulmonary toxicity, such as pulmonary fibrosis, organizing pneumonia (e.g., obliterative bronchiolitis), pneumoconiosis, drug-related pneumonia, idiopathic pneumonia, or subjects with active pneumonia or severe lung function impairment shown by chest CT during screening; active tuberculosis;
4. Presence of active autoimmune diseases or a history of autoimmune diseases that may relapse [including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (patients controlled only by hormone replacement therapy can be included)]; patients with skin diseases that do not require systemic treatment, such as vitiligo, psoriasis, alopecia, controlled type 1 diabetes mellitus treated with insulin, or patients with asthma who have completely resolved in childhood and require no intervention as adults can be included; patients with asthma requiring bronchodilators for medical intervention cannot be included;
5. Within 2 weeks before the start of the study, use of immunosuppressants or systemic hormone therapy to achieve immunosuppression (dose >10mg/day prednisone or other equivalent glucocorticoids);
6. Patients with active infections, with unexplained fever ≥38.5°C within 1 week before the start of the study, or with a baseline white blood cell count >15×10^9/L;
7. Patients with congenital or acquired immune deficiency (e.g., HIV infection);
8. Within 4 weeks before the first dose, received or planned to receive live or attenuated live vaccines during the study;
9. Within 6 months before the start of the study, significant clinical bleeding symptoms or a clear bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, or vasculitis, etc. If positive for occult blood in stool at baseline, it can be retested; if still positive after retesting, endoscopy is required;
10. Known existing hereditary or acquired bleeding disorders (e.g., hemophilia patients), coagulation disorders, thrombocytopenia, etc.); currently receiving full-dose oral or injected anticoagulants or thrombolytics for therapeutic purposes (prophylactic use of low-dose aspirin is allowed, etc.);
11. Within 6 months before the start of the study, arterial thromboembolic events, such as cerebrovascular accidents (including transient ischemic attacks, intracerebral hemorrhage, cerebral infarction), CTCAE grade 3 or higher deep vein thrombosis, pulmonary embolism, etc;
12. Uncontrolled heart clinical symptoms or diseases, such as: (1) New York Heart Association (NYHA) standard II or higher heart failure or echocardiography: LVEF (left ventricular ejection fraction) <50%; (2) unstable angina pectoris; (3) myocardial infarction within 1 year before treatment; (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention; (5) QTc >450ms (men); QTc >470ms (women) (QTc interval calculated using the Fridericia formula: if QTc is abnormal, it can be continuously measured for 3 times at intervals of 2 minutes and the average value is taken);
13. Hypertension that cannot be well controlled with antihypertensive medication (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg) (based on the average of blood pressure readings from ≥2 measurements); previous history of hypertensive emergencies or hypertensive encephalopathy is allowed;
14. Within 6 months before the start of the study, the occurrence of major vascular diseases (e.g., aortic aneurysms requiring surgical repair or recent peripheral arterial thrombosis);
15. Severe, unhealed, or open wounds, as well as active ulcerations or untreated fractures;
16. Within 4 weeks before the start of the study, received major surgery treatment (excluding diagnostic procedures) or expect to undergo major surgery during the study period;
17. Unable to swallow pills, malabsorption syndrome, or any condition that affects gastrointestinal absorption;
18. Within 6 months before the start of the study, experienced intestinal obstruction and/or had clinical signs or symptoms of gastrointestinal obstruction, including incomplete obstruction related to the original disease or requiring routine parenteral hydration, parenteral nutrition, or tube feeding. If patients with incomplete obstruction/obstruction syndrome/intestinal obstruction signs/symptoms at the time of initial diagnosis received definitive (surgical) treatment to resolve symptoms, they may be eligible for inclusion in the study;
19. Within 2 weeks before the start of the study, the use of strong CYP3A4/CYP2C1 inducers including rifampicin (and its analogues) and St. John's wort, or strong CYP3A4/CYP2C19 inhibitors;
20. Subjects who have received other neoantigen vaccines, or are allergic to any chemotherapy drugs, anti-angiogenic targeted drugs, or excipients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) and Treatment-Related Adverse events (TRAEs), Serious adverse events (SAEs), and grade 3 or higher TRAEs. | Up to 12 weeks after the last use of the study drug
  Safety parameters in this study include clinical symptoms, vital signs, physical examinations, laboratory tests (complete blood count, urinalysis, blood chemistry, coagulation function, etc.). Adverse events (AEs) observed are evaluated according to the NCI-CTCAE version 5.0, including type, incidence, severity, onset and end time, whether they are serious adverse events, and their relationship to the investigational drug.

SECONDARY OUTCOMES:
1 year Overall Survival (OS) rate | up to 1 year
  The percentage of patients who are still alive one year after the start of the study.
Recurrence-free survival (RFS) | up to 2 years
  Recurrence-free survival (RFS) is defined as the time from initiation of treatment with the first dose to the first documented recurrence (according to RECIST 1.1 criteria) or until the patient's death from any cause, whichever occurs first.

OTHER OUTCOMES:
Biomarker analysis (changes in immune cells and regulating immune-related molecules and immune-related indicators in patients before and after treatment) | Up to 2 years
  Assess the effects of new antigen vaccines on activating immune cells and regulating immune-related molecules, as well as changes in immune-related indicators in patients before and after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Mengchao Hepatobiliary Hospital, Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No